CLINICAL TRIAL: NCT04769687
Title: Symbiotics and Systemic Inflammation in Chronic Kidney Disease
Acronym: SISMIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: API/2016/76 2019-A00850-57
Record Dates: First submitted 2020-09-04; First posted 2021-02-24 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Chronic Renal Failure; Diabete Type 2; Systemic Inflammation
Keywords: Inflammation; Chronic renal failure; Symbiotic
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetes Mellitus, Type 2; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized, non-comparative 2: 1 phase 2 study (symbiotic vs placebo) aimed at evaluating the efficacy of the use of symbiotics in reducing chronic inflammation observed in chronic renal failure.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symbiotic Treatment : probiotic Vivomixx® + prebiotic Orafti®Synergy1 (Experimental): The prebiotic, Orafti®Synergy1, is made from a volume-to-volume mixture of oligofructoses and Raftiline HP. Orafti®Synergy1 is a slightly sweet white powder packaged in 5 g sachets that can be administered orally. The dose used is 2 sachets per day (morning and evening) for 8 weeks (56 days).
  The probiotic, Vivomixx®, consists of 4 strains of Lactobacillus (L. casei, L. plantarum, L. acidophilus and L. delbrueckii subsp. Bulgaricus) from 3 strains of Bifidobacterium (B. longum, B. breve, and B. infantis) and a strain of streptococcus (S. salivarius subsp thermophilus). Vivomixx® is in powder form packaged in sachets of 4.5.1011 bacteria which can be administered orally. The dose used is 2 sachets per day (morning and evening) for 8 weeks (56 days).
  For the study, the symbiotics will be packaged by the probiotic manufacturer in the same sachet (at the same doses as mentioned above) whether for the symbiotics or for the placebo.
  Interventions: Biological: probiotic Vivomixx®; Biological: prebiotic Orafti®Synergy1
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: probiotic Vivomixx® — Vivomixx® is in powder form packaged in sachets of 4.5.1011 bacteria. The dose used is 2 sachets per day (morning and evening) for 8 weeks (56 days). For the study, the symbiotics will be packaged in the same sachet at the same doses as mentioned above.
  Arms: Symbiotic Treatment : probiotic Vivomixx® + prebiotic Orafti®Synergy1
Biological: prebiotic Orafti®Synergy1 — Orafti®Synergy1 is a slightly sweet white powder packaged in 5 g sachets. The dose used is 2 sachets per day (morning and evening) for 8 weeks (56 days).
  Arms: Symbiotic Treatment : probiotic Vivomixx® + prebiotic Orafti®Synergy1
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Main objective: To assess the effectiveness of treatment with symbiotics on the chronic systemic inflammation observed in chronic renal failure 4 months after the start of treatment.

DETAILED DESCRIPTION:
During a consultation in the nephrology departments : the study will be presented to the patient and the information leaflet will be given to him.

During a subsequent visit, after checking the level of serum CRP and obtaining the consent of the investigating physician, a blood test will be taken to assess the intestinal permeability and the inflammatory state. A health-related quality of life (SF-36) and frailty questionnaire (previous questionnaire, MNA questionnaire; Mini Nutritional Assessment - Short Form and physical activity question) will be completed by the patient. Two faecal sampling kits (one for D0 and one for M2) will be distributed to patients.

During the D0 visit, patients will be randomized into two arms. Both arms will receive the same dietary advice. The intervention group will receive symbiotics (prebiotics: Orafti®Synergy1 and probiotics: Vivomixx®) for 8 weeks against a placebo in the control group. The treatment will begin after the collection of the first stools (kit J0).

At the end of the treatment (M2 or 56 days later), a new blood sample will be taken. Two other blood samples will be taken 4 months and 6 months after the start of treatment. Patients will also provide a faecal sample and complete the various questionnaires at the end of treatment (M2), 2 months after (M4) and 4 months after (M6) treatment.

The study will have no influence on the management of the patient. It does not require any additional consultation or any particular biological assessment other than that described. Treatments should not be influenced by the study. The samples will be processed without knowledge of the initial characteristics of the patients, nor of their evolution.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 80 inclusive
* Women who have been menopausal for at least 24 months, surgically sterilized, or, for women of childbearing potential, use an effective method of contraception (oral contraceptives, contraceptive injections, intrauterine devices, double-barrier method, contraceptive patches)
* Signature of the informed consent to participate indicating that the subject has understood the purpose and the procedures required by the study and that he agrees to participate in the study and to comply with the requirements and restrictions inherent in this study
* Affiliation to a French social security scheme or beneficiary of such a scheme.
* Patient with type II diabetes
* Creatinine clearance less than 45 ml / min / 1.73m²
* Serum CRPus level greater than 6 mg / l, evaluated twice from 15 days to 3 months apart
* Patient not opposed to the conservation of biological samples for scientific research purposes.

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate with the study and / or weak cooperation anticipated by the investigator
* Subject without health insurance
* Pregnant woman
* Subject being in the period of exclusion from another study or provided for by the "national file of volunteers".
* Infectious episode with need for hospitalization less than 1 month old.
* Active infection with hepatitis B and / or C virus.
* Active or non-progressive infection with HIV.
* Antibiotic therapy in the previous 3 months.
* Anti-inflammatory treatment.
* History of colectomy.
* All chronic digestive pathologies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-11-21 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
inflammation | 4 months
  change in inflammation estimated by the serum CRP concentration <6 mg / L

SECONDARY OUTCOMES:
inflammatory cytokines 1 | At 2, 4 and 6 months after the start of treatment.
  variation of IL-6
inflammatory cytokines 2 | At 2, 4 and 6 months after the start of treatment.
  variation of IL-1β
inflammatory cytokines 3 | At 2, 4 and 6 months after the start of treatment.
  variation of TNF-α
inflammatory cytokines 4 | At 2, 4 and 6 months after the start of treatment.
  variation of IL-10
inflammatory cytokines 5 | At 2, 4 and 6 months after the start of treatment.
  variation of IL-8
inflammatory cytokines 6 | At 2, 4 and 6 months after the start of treatment.
  variation of IFNγ
inflammatory circulating monocytes | At 2, 4 and 6 months after the start of treatment.
  variation
intestinal microbial metabolome | At 2, 4 and 6 months after the start of treatment.
  modification of the intestinal microbial metabolome (Nuclear magnetic resonance)
intestinal membrane permeability | At 2, 4 and 6 months after the start of treatment.
  modification of LPS
bacterial translocation 1 | At 2, 4 and 6 months after the start of treatment.
  modification of CD14s
bacterial translocation 2 | At 2, 4 and 6 months after the start of treatment.
  modification of iFABP
health-related quality of life | At 2, 4 and 6 months after the start of treatment.
  SF-36 Health Survey (Short Form) The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
fragility | At 2, 4 and 6 months after the start of treatment.
  fragility (= 3 of the following 5 criteria: undernutrition, grip strength and walking speed, assessed exhaustion and physical activity)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No
Individual data can be provided on request after validation by the competent regulatory authorities.